CLINICAL TRIAL: NCT00002336
Title: A Prospective, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study of the Safety and Efficacy of Clarithromycin for the Prevention of Disseminated Mycobacterium Avium Complex (MAC) Infection in HIV-Infected Patients With CD4 Counts <= 100 Cells/mm3
Brief Title: The Safety and Effectiveness of Clarithromycin in the Prevention of Mycobacterium Avium Complex (MAC) Infection in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 124A; M91-561
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2009-02

CONDITIONS: Mycobacterium Avium-intracellular Infection; HIV Infections
Keywords: Mycobacterium avium-intracellular Infection; Acquired Immunodeficiency Syndrome; Clarithromycin
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Clarithromycin

INTERVENTIONS:
Drug: Clarithromycin

SUMMARY:
To determine whether clarithromycin is safe and effective in preventing disseminated Mycobacterium avium Complex in HIV-infected patients with CD4 counts <= 100 cells/mm3.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV infection.
* CD4 count <= 100 cells/mm3.
* No evidence of MAC.
* Life expectancy of at least 6 months.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Certain restricted drugs (details not available).

Patients with the following prior conditions are excluded:

History of allergy or hypersensitivity to macrolides. Active substance abuse or other conditions that would affect study compliance.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-11; Primary Completion 1994-11 (Actual); Study Completion 1994-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (22):
  - Univ of Arizona / Health Science Ctr, Tucson, Arizona
  - California Med Research Group, Fresno, California
  - HIV Research Group, San Diego, California
  - Saint Francis Mem Hosp, San Francisco, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - TheraFirst Med Ctrs Inc, Fort Lauderdale, Florida
  - Dr Nelson Zide, Hollywood, Florida
  - Infectious Disease Research Institute Inc, Tampa, Florida
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Saint Vincent's Hosp and Med Ctr, New York, New York
  - SUNY / Health Sciences Ctr at Syracuse, Syracuse, New York
  - New York Med College / Westchester County Med Ctr, Valhalla, New York
  - Nalle Clinic, Charlotte, North Carolina
  - Westover Heights Clinic, Portland, Oregon
  - Univ of Tennessee, Memphis, Tennessee
  - Vanderbilt Univ, Nashville, Tennessee
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Houston Veterans Administration Med Ctr, Houston, Texas
  - Audie L Murphy Veterans Administration Hosp, San Antonio, Texas
  - Salem Veterans Administration Med Ctr, Salem, Virginia
  - Dr Alan D Tice / Infections Ltd, Tacoma, Washington

REFERENCES:
- [Background] Pierce M, Crampton S, Henry D, Heifets L, LaMarca A, Montecalvo M, Wormser GP, Jablonowski H, Jemsek J, Cynamon M, Yangco BG, Notario G, Craft JC. A randomized trial of clarithromycin as prophylaxis against disseminated Mycobacterium avium complex infection in patients with advanced acquired immunodeficiency syndrome. N Engl J Med. 1996 Aug 8;335(6):384-91. doi: 10.1056/NEJM199608083350603. PMID 8663871